CLINICAL TRIAL: NCT01516866
Title: NaF PET/CT Repeatability, Responsiveness, and Response Assessment in Patients With Metastatic Castrate-resistant Prostate Cancer to Bone Treated With Either an Antimicrotubule Directed Agent or Androgen Receptor (AR)-Directed Therapies
Brief Title: Sodium Fluoride (NaF) Positron Emission Tomography/Computed Tomography (PET/CT) in Patients With Metastatic Castrate-resistant Prostate Cancer (CRPC) With Microtubule Directed Chemo or AR-directed Therapy
Acronym: NaFl PET/CT
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: CO11811; 2011-0397 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison)
Record Dates: First submitted 2011-11-28; First posted 2012-01-25 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2018-04

CONDITIONS: Prostate Cancer
Keywords: Androgen receptor-directed therapy; NaF PET/CT; antimicrotubule directed chemotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sodium Fluoride; Magnetic Resonance Spectroscopy; X-Rays

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cohort A: Microtubule directed chemotherapy treatment: Subjects receiving antimicrotubule chemotherapy-based treatment will have NaF PET/CT scans at baseline and again after 8 weeks of starting treatment. A subset of subjects will have a second NaF PET/CT scan at baseline 1-8 days after the first baseline scan.
  Interventions: Procedure: Sodium Fluoride (NaF) Positron Emission Tomography/Computed Tomography (PET/CT) imaging
- Cohort B: AR-directed therapy: Subjects receiving AR-directed therapy will undergo a baseline NaF PET/CT scan at baseline and again after having been on treatment for 6 weeks and again at 12 weeks. A subset of subjects will also undergo a second baseline NaF PET/CT scan 1-8 days after the first baseline scan.
  Interventions: Procedure: Sodium Fluoride (NaF) Positron Emission Tomography/Computed Tomography (PET/CT) imaging

INTERVENTIONS:
Procedure: Sodium Fluoride (NaF) Positron Emission Tomography/Computed Tomography (PET/CT) imaging — Subjects who will be enrolled will be those who will be starting treatment (as part of standard of care or as part of another trial) with either a microtubule directed chemotherapy regimen (cohort A), or AR-directed therapy (cohort B). All subjects will have a baseline NaF PET/CT scan (baseline #1), performed within days prior to starting either chemotherapy or AR-directed therapy. A subset of subjects (up to 20 subjects per site, 60 total) will undergo a second NaF PET/CT scan (baseline #2) within 1-8 days of the initial scan to determine repeatability of NaF PET/CT scanning. Subjects in cohort A will undergo another NaF PET/CT scan at week 8 (+/- 1 week). Subjects in cohort B will undergo two additional NaF PET/CT scans at weeks 6 and 12 (+/- 1 week).

SUMMARY:
The purpose of this research study is to evaluate a newer imaging technique, called 18F-Sodium Fluoride (NaF) positron emission tomography (PET). NaF is a tracer (dye) that is very sensitive for changes in bone. By using this tracer with positron emission tomography/computed tomography (PET/CT) imaging, our ability to evaluate and measure changes in bone lesions could be greatly improved.

DETAILED DESCRIPTION:
The study will look at how repeatable the NaF PET scans are before treatment. Scans will also be performed after standard chemotherapy or hormone-directed treatment. This will allow evaluation of how the NaF PET scans change with the chemotherapy or hormone-directed therapy. In addition, NaF PET scans will be compared with standard computed tomography (CT) and bone scans, as well as prostate specific antigen (PSA). This information could be used to develop better ways to measure prostate cancer bone lesions. In turn, this could be used to better evaluate treatment effects of standard chemotherapy and other new drugs being developed to treat prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Identifiable prostate cancer-related bone metastases on bone scan in the spine, pelvis or other bone
* Patients must be starting a microtubule directed chemotherapy regimen for metastatic castrate-resistant prostate cancer OR
* Patients must be starting a AR-directed regimen (e.g. Abiraterone, MDV-3100, TAK-700, etc) for treatment of metastatic castrate-resistant prostate

Exclusion Criteria:

* Concurrent treatment with any other agent that is being used with the expressed purpose of treating of prostate cancer outside of the planned treatment regimen
* Patients who have received radiotherapy less than 4 weeks prior to registration.
* Patients who have received prior Strontium-89, Samarium-153, or other radioisotope.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sodium fluoride F-18 (NaF).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
The repeatability of NaF PET/CT imaging for evaluating bone metastases in patients with metastatic castrate-resistant prostate cancer. | 2 years
  NaF PET/CT scan will be performed within 14 days prior to starting chemotherapy (antimicrotubule directed chemotherapy) or hormone-directed therapy (baseline #1). A portion of subjects (up to 20 subjects at each site, 60 subjects total) will have a second NaF PET/CT scan performed (baseline #2) within 1-8 days of the initial scan to see if measurements repeated over a short period of time are similar.

SECONDARY OUTCOMES:
Evaluate changes on NaF PET/CT images in response to chemotherapy (antimicrotubule directed chemotherapy) or androgen receptor (AR)-directed therapy. | 2 years
  All subjects will undergo NaF PET/CT scanning at baseline and again either 8 weeks after starting treatment with antimicrotubule chemotherapy based treatment (Cohort A) OR at both 6 weeks and 12 weeks after starting AR-directed treatment (Cohort B).
Prostate Specific Antigen (PSA) response | 2 years
  Results from the NaF PET/CT scans will be compared with PSA and bone scan and CT scan results.
Response Evaluation Criteria in Solid Tumors (RECIST) response | 2 years
Radiographic progression free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Liu, MD, Principal Investigator — University of Wisconsin, Madison; Robert Jeraj, Ph.D., Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - National Cancer Institute, Bethesda, Maryland
  - Memorial Sloan Kettering, New York, New York
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/